CLINICAL TRIAL: NCT06241001
Title: Effect of Eccentric Streching vs IASTM of Gastrocnemius and Soleus Muscles in Athletes With Ankle Sprain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RiphahIU Asim
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Ankle Sprains
Keywords: Soleus; Gastrocnemius; eccentric; IASTM
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eccentric streching (Experimental): Group A will receive eccentric stretching for ankle sprain
  Interventions: Other: eccentric streching
- IASTM (Active Comparator): Group B will only receive IASTM.
  Interventions: Other: IASTM

INTERVENTIONS:
Other: eccentric streching — The player will lift up one leg from starting position so he stands on his to-be-trained leg. For performing eccentric exercises of the gastrocnemius muscles, the player will lower his heel until he will feel a slight stretch, while keeping his knee extended
  Arms: Eccentric streching
Other: IASTM — Specially designed tools are used to apply longitudinal pressure along muscle fibers, and treatment usually includes applying to more than the tissues in the isolated location of the pain
  Arms: IASTM

SUMMARY:
The primary objective within the current study is to compare the acute and chronic effects of eccentric training and IASTM on the dorsiflexion ROM. To reduce the risk of Achilles tendinopathy, stretching and eccentric (lengthening) exercises are postulated to improve ankle dorsiflexion. An eccentric exercise lengthens an active muscle while it is under load. Consequently, eccentric calf muscle exercises can also increase ankle dorsiflexion through an increase in calf muscle strength. For the above mentioned reasons, a combination of stretching exercises and eccentric (lengthening) exercises are suggested as preventive intervention to increase ankle dorsiflexion. The biggest goal of IASTM is to remove scar tissues and facilitate a return to normal function following soft tissue recovery. These Techniques, eccentric stretching and IASTM works towards bringing back the normal range of motion and strength, allowing individuals to regain mobility and return to their usual activities and we will find out the better option from these.

DETAILED DESCRIPTION:
Ankle sprain is a traumatic injury that occurs to one or more of lateral ankle ligaments: anterior talofibular ligament, posterior talofibular ligament and calcaneofibular ligament. Ankle sprains are one of the most common musculoskeletal injuries. The ankle is the second most commonly injured body part during sports, with ankle sprains being the most common ankle injury. Instrument-Assisted Soft Tissue Mobilization (IASTM) is a type of soft tissue mobilization that uses rigid devices to increase the examination and treatment of soft tissues. According to recent studies, Instrument-Assisted Soft Tissue Mobilization (IASTM) is a new and highly trained myofascial technique that has gained favor in modern decades for treating soft-tissue ailments. To reduce the risk of Achilles tendinopathy, stretching and eccentric (lengthening) exercises are postulated to improve ankle dorsiflexion. An eccentric exercise lengthens an active muscle while it is under load.

Consequently, eccentric calf muscle exercises can also increase ankle dorsiflexion through an increase in calf muscle strength. For the above mentioned reasons, a combination of stretching exercises and eccentric (lengthening) exercises are suggested as preventive intervention to increase ankle dorsiflexion. Eccentric training is an alternative modality that also shows promise for inducing chronic improvement in ROM. In past years there has been different protocols to treat ankle sprain but this study will contribute to more effective method of treating ankle sprain, improving their recovery and also reducing the risk of re-injury. This study will potentially reduce healthcare costs associated with rehabilitation or the need of additional interventions. This study will have fast and more effective rehabilitation method which can boost the athlete performance, making it the treatment of choice for both athletes and sports teams.

ELIGIBILITY:
Inclusion Criteria:

Age 18 and above Both genders Ankle sprain acute and Sub acute

Exclusion Criteria:

Acute fracture to lower extremity Arthritis patients Any other trauma or injury to the lower extremity

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Foot and Ankle Ability Measure (FAAM) | four weeks
  The Foot and Ankle Ability Measure (FAAM) is a self-report outcome instrument developed to assess physical function for individuals with foot and ankle related impairments
NPRS | four weeks
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain)
Goniometer | four weeks
  A goniometer is a device used in physical therapy to measure a joint's range of motion (ROM).

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Wasay Nafe, MS-SPT, Principal Investigator — Riphah International University
Locations (1):
- Railway General Hospital, Rawalpindi, Pakistan

IPD SHARING:
Plan to Share IPD: No